CLINICAL TRIAL: NCT00904176
Title: Study of the Effect of Dapagliflozin on the Pharmacokinetics of Warfarin or Digoxin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MB102-058
Record Dates: First submitted 2009-05-18; First posted 2009-05-19 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Warfarin; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dapagliflozin + Warfarin (Active Comparator)
  Interventions: Drug: Dapagliflozin; Drug: Warfarin
- Warfarin (Active Comparator)
  Interventions: Drug: Warfarin
- Dapagliflozin + Digoxin (Active Comparator)
  Interventions: Drug: Dapagliflozin; Drug: Digoxin
- Digoxin (Active Comparator)
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 20 mg, followed by 10 mg, Single Dose
  Arms: Dapagliflozin + Digoxin; Dapagliflozin + Warfarin
Drug: Warfarin — Tablets, Oral, 25 mg, Single Dose
  Other Names: Coumadin
  Arms: Dapagliflozin + Warfarin; Warfarin
Drug: Digoxin — Tablets, Oral, 0.25, Single Dose
  Other Names: Lanoxin
  Arms: Dapagliflozin + Digoxin; Digoxin

SUMMARY:
The purpose of this study is determine that Dapagliflozin has no effect on the pharmacokinetics (PK) or pharmacodynamics (PD) of warfarin when dapagliflozin is coadministered with warfarin. Also, that Dapagliflozin has no effect on the PK of digoxin when dapagliflozin is coadministered with digoxin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m², inclusive. BMI = weight (kg)/ [height (m)]²
* Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) and men, ages 18 to 45

Exclusion Criteria:

* WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal
* Any significant acute or chronic medical illness or relevant trauma (e.g. history of chronic hypertension, bacterial endocarditis, hemorrhagic stroke, motor vehicle accident resulting in significant head trauma or internal injuries)
* History of important arrhythmias as determined by the Investigator, including but not limited to ventricular fibrillation, ventricular tachycardia, A-V block, Wolff-Parkinson-White Syndrome, and sinus bradycardia (defined in this study as heart rate < 50 bpm based on vital signs and ECG performed within 21 days of Study Day 1)
* History or evidence of abnormal bleeding or coagulation disorder (e.g., history of prolonged bleeding during dental procedures, pregnancy delivery, previous surgery or injury) and/or having a first degree relative under 50 years of age with a history of abnormal bleeding or coagulation disorder per patient's report
* History of unexplained syncope
* Presence of external hemorrhoids with signs of rectal bleeding on physical exam
* Positive fecal occult blood (FOB), using the Hemoccult Sensa® assay (or equivalent), or hematuria (more than trace), unless deemed not clinically significant by the Investigator and Medical Monitor at screening or dosing
* Platelet count < 150,000 cells/µL at screening or dosing
* INR or aPTT values above the upper limit of normal (ULN) at screening or dosing
* Hemoglobin or hematocrit < LLN at screening or dosing
* Abnormal urinalysis at screening or dosing (repeat urinalysis may be allowed for positive hematuria in women)
* Glucosuria at screening or dosing
* Abnormal liver functions tests (ALT, AST or total bilirubin > 10% above ULN) at screening or dosing
* History of diabetes mellitus
* History of heart failure
* History of renal insufficiency
* History of recurrent (defined as 3 occurrences per year) or recent vulvovaginal mycotic infections
* Positive urine screen for drugs of abuse either at screening or before dosing
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or HIV-1, -2 antibody
* Protein C or Protein S deficiency
* History of allergy to SGLT2 inhibitors or related compounds
* History of allergy to warfarin or related compounds
* History of allergy to digoxin or related compounds
* Prior exposure to dapagliflozin within 3 months of Day -1
* Exposure to any investigational drug or placebo within 4 weeks of Day -1
* Use of any prescription drugs within or over-the-counter acid controllers or vitamin K containing products within 4 weeks prior to study drug administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Exposure to the investigational drug will be measured to compare with and without the co-administration of other drugs | 216 hours post-dose

SECONDARY OUTCOMES:
To assess the effect of dapagliflozin on the PK of R-warfarin, when warfarin and dapagliflozin are coadministered in healthy subjects (Cohort 1) | 16 time points
To assess the safety and tolerability of the combination of dapagliflozin with warfarin, and the combination of dapagliflozin with digoxin in healthy subjects | 16 time points

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Pra International, Lenexa, Kansas, United States

REFERENCES:
- See also: MB102-058_redacted _CSR _synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3648&filename=MB102-058_redacted%20_CSR%20_synopsis.pdf